CLINICAL TRIAL: NCT01679301
Title: Evaluation of Sleep Mode Within the Respironics SimplyGo Portable Oxygen Concentrator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HRC-1216-SimGoSleep-SS
Record Dates: First submitted 2012-08-24; First posted 2012-09-06 (Estimated); Results first posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Lung Disease
Keywords: oxygen
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous dose (Active Comparator): Users will be randomized to either receive oxygen via continuous dose oxygen or pulsed dose ('sleep' mode) for the first part of the night and will switch for the second part of the night using the SimplyGo Portable Oxygen Concentrator.
  Interventions: Device: Continuous Dose
- Pulse dose ('sleep mode') (Experimental): Users will be randomized to either receive oxygen via continuous dose oxygen or pulsed dose ('sleep' mode) for the first part of the night and will switch for the second part of the night using the SimplyGo Portable Oxygen Concentrator
  Interventions: Device: Pulse Dose (Sleep Mode)

INTERVENTIONS:
Device: Pulse Dose (Sleep Mode) — SimplyGo Portable Oxygen Concentrator has two different modes of use 'Sleep Mode', or pulsed oxygen and continuous dose.
  Arms: Pulse dose ('sleep mode')
Device: Continuous Dose — SimplyGo Portable Oxygen Concentrator has two different modes of use 'Sleep Mode', or pulsed oxygen and continuous dose.
  Arms: Continuous dose

SUMMARY:
The SimplyGo Study is a single site, cross-over study which aims to enroll a maximum of 30 participants (to allow for 20 completed data sets) with a prescription for nocturnal oxygen, and meeting all eligibility criteria.

DETAILED DESCRIPTION:
All participants will undergo a single night polysomnography testing in a sleep lab while they're oxygen saturation (SpO2) is monitored. The study has a cross-over design, in which participants will receive their oxygen prescription in two different modes at different times during the night. The assignment (sleep vs. continuous mode) to which participants will initiate the night will be randomized, and all participants will utilize each of the two modes during the study. The hypothesis of this study is that there will not be a significant difference in SpO2 for participants while they use the SimplyGo Portable Oxygen Concentrator, set in 'Sleep Mode', or pulsed oxygen flow, as compared to their SpO2 while on continuous flow oxygen during sleep during the course of the one night sleep study.

ELIGIBILITY:
Inclusion Criteria

1. Males and Females, ages 21-80
2. Current prescription for supplemental oxygen at night; Can be pulsed dose or continuous
3. Willing and able to provide informed consent

Exclusion Criteria

1. Medically unstable participants per discretion of the principal investigator
2. Diagnosis of sleep apnea, per chart review, self report or rated high risk based on the Berlin Questionnaire
3. Participants unable or unwilling to spend one night in a sleep lab
4. Nocturnal oxygen requirements > 5 liters per minute
5. Currently employed by a manufacturer of respiratory products or family member employed by a manufacturer of respiratory products
6. Employee or family member that is affiliated with Philips

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sukhdev Grover, MD, Principal Investigator — Medical Director, Sukhdev Grover and Associates
Locations (1):
- Sukhdev Grover and Associates, Monroeville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants: All Participants enrolled in the study
- Continuous Dose Then Pulse Dose ('Sleep Mode'): Users will be randomized to either receive oxygen via continuous dose oxygen or pulsed dose ('sleep' mode) for the first part of the night and will switch for the second part of the night using the SimplyGo Portable Oxygen Concentrator.
  Continuous Dose: SimplyGo Portable Oxygen Concentrator has two different modes of use 'Sleep Mode', or pulsed oxygen and continuous dose.
- Pulse Dose ('Sleep Mode') Then Continuous Dose: Users will be randomized to either receive oxygen via continuous dose oxygen or pulsed dose ('sleep' mode) for the first part of the night and will switch for the second part of the night using the SimplyGo Portable Oxygen Concentrator Pulse Dose (Sleep Mode): SimplyGo Portable Oxygen Concentrator has two different modes of use 'Sleep Mode', or pulsed oxygen and continuous dose.
Period: Screening Period
Arm/Group | Participants | Continuous Dose Then Pulse Dose ('Sleep Mode') | Pulse Dose ('Sleep Mode') Then Continuous Dose
Started | 11 | 0 | 0
Completed | 8 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — screen failure | 3 | 0 | 0
Period: Study Period
Arm/Group | Participants | Continuous Dose Then Pulse Dose ('Sleep Mode') | Pulse Dose ('Sleep Mode') Then Continuous Dose
Started | 0 | 4 | 4
Completed | 0 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 11 participants were consented for the trial, after consent 3 were found to be not eligible and 8 continued into the trial and completed.
Arm/Group | Participants
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.76 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.25 (9.8)

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Saturation Values Obtained From Pulse Oximetry
Description: A comparison of the average oxygen saturation values obtained via pulse oximetry during continous flow oxygen versus 'sleep' mode while sleeping
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation (SpO2)
Arm/Group | Continuous Dose | Pulse Dose ('Sleep Mode')
Number analyzed (Participants) | 8 | 8
percentage of oxygen saturation (SpO2)
  Oxygen Saturation (SpO2) while Awake | 97.6 (1.14) | 95.8 (1.92)
  SpO2 while in non rapid eye movement sleep (NREM) | 97 (2.45) | 96 (2.1)
  SpO2 while in rapid eye movement sleep (REM) | 100 (0) | 97.5 (2.38)
  SpO2 over while in bed (TIB (time in bed)) | 97 (2.45) | 96.2 (2.23)

ADVERSE EVENTS:
Time Frame: 1 night
Description: 8 participants completed one overnight visit in the lab, during the night participants were monitored for adverse events.
Groups:
- Continuous Dose: Users will be randomized to either receive oxygen via continuous dose oxygen or pulsed dose ('sleep' mode) for the first part of the night and will switch for the second part of the night using the SimplyGo Portable Oxygen Concentrator.
  Dose: SimplyGo Portable Oxygen Concentrator has two different modes of use 'Sleep Mode', or pulsed oxygen and continuous dose
Arm/Group | Continuous Dose | Pulse Dose ('Sleep Mode')
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No